CLINICAL TRIAL: NCT03665974
Title: Lower Vitamin D Levels During Second Trimester Are Associated With Developing Gestational Diabetes Mellitus: an Observational Cross-sectional Study
Brief Title: The Relation Between Vitamin D and Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, F. Gülhan Samur, Professor doctor, Hacettepe University
Other Study IDs: Hacettepe University Nutrition
Record Dates: First submitted 2018-09-06; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Deficiency, Vitamin D; Diabetes, Gestational
Keywords: Pregnancy, deficinecy, vitamin D, diabetes, gestational
MeSH Terms: conditions — Vitamin D Deficiency; Diabetes, Gestational; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with gestational diabetes mellitus: GDM screening at this hospital involves a two-step procedure. The diagnosis of GDM was confirmed if at least 2 of 4 glucose levels exceed based on Carpenter-Coustan criteria: fasting ≥ 95 mg/dL (5.3 mmol/L), 1 hour ≥ 180 mg/dL ( 10.0 mmol/L), 2 hour ≥ 155 mg/dL (8.6 mmol/L), and 3 hour ≥ 140 mg/dL (7.8 mmol/L).
- Women non gestational diabetes mellitus: Women with normal serum glucose levels ≤129 mg/dL (7.2 mmol/L) after GCT.

SUMMARY:
Gestational diabetes mellitus (GDM) is defined as any degree of glucose intolerance with the onset or first recognition during pregnancy. The prevalence of GDM varies from 1-14% due to its variability worldwide, depending on the ethnicity, race, and the diagnostic criteria being applied by each country. In addition to this, approximately 7% of all pregnancies are affected by GDM, ending up more than 200,000 women with GDM per year. A recent study of literature research indicated that Middle East and North Africa had the highest prevalence (median, 12.9%) while Europe had the lowest prevalence (median, 5.8%) in the world. In Turkey the prevalence of GDM ranges between 4-10%, based on the reports in different studies.

As a growing health concern, GDM has been associated with short and long-term detrimental health outcomes for women and their offspring. Maternal adverse effects of GDM are preeclampsia, elevated risk of development of hypertension, type 2 diabetes mellitus (T2DM), urinary tract infection and comorbidities following delivery. Macrosomia, neonatal jaundice, birth trauma, respiratory distress syndrome, hypoglycemia are included in short term consequence for the neonates whereas risk for development of impaired glucose tolerance, T2DM, obesity, vascular disorders are long term adverse effects on infant's health.

The known risk factors for GDM include family history of T2DM, maternal overweight and obesity, advanced maternal age, history of GDM, having macrosomic infant previously, prior fetal death, and race/ethnicity. In addition to these risk factors, recent studies have been suggested that maternal vitamin D deficiency may be associated with a higher risk of GDM.

Vitamin D deficiency during the pregnancy has been associated with adverse outcomes for the pregnant women, such as gestational diabetes mellitus, urinary tract infection, preeclampsia, caesarean section during labour [25]. Furthermore, infants born to mothers with lower vitamin D levels have been found to be associated with elevated risk of small for gestational age, low birth weight in the neonatal period, increased risk for cardiovascular disease, respiratory illnesses, type 2 diabetes mellitus in childhood and adulthood.

The aim of this study was to compare the serum 25(OH)D levels of women with and without gestational diabetes mellitus (GDM) and identify the serum 25(OH)D level associated with GDM during pregnancy.

DETAILED DESCRIPTION:
In this observational cross-sectional study, 40 women with GDM and 40 healthy pregnant between 20-40 years in age, in their 24-28th gestational week applied to Gulhane Education and Research Hospital (Ankara, Turkey) were recruited between January 2014 to March 2014. Inclusion criteria were singleton pregnancy, aged 20-40 years, gestational age 24-28 weeks, non-history of acute or chronic diseases. The exclusion criteria included alcohol using, smoking, history of GDM, diagnosed with type 1 and 2 diabetes mellitus, preeclampsia, polycystic ovary syndrome, thyroid and parathyroid disease, metabolic bone disease, kidney disease, abnormal liver function, multiple pregnancy, or women receiving drugs related to calcium and vitamin D metabolism (with the exception of routine vitamin supplements prescribed during pregnancy). We randomly selected the 40 pregnant women diagnosed GDM by two-step procedure based on Carpenter-Coustan criteria. Women with GDM did not receive any type of the medications such as insulin or medical nutrition therapy. We also randomly selected 40 healthy pregnant women with normal serum glucose levels in the same period. This study must recruit 40 women for each group to have 80% study power with 5% type I error level to detect a clinically significant difference.

The study was approved by the ethic committee of Gulhane Education and Research Hospital, Ankara, Turkey with the number 50687469-1491-2721-13/1648.4-2882. Before commencing the research, not only women got clued in information about the study procedure and objective but also a written informed consent was obtained from all participants.

GDM screening at this hospital involves a two-step procedure. At the outset, 50 g 1 hour glucose challenge test (GCT) was used to screen for GDM at 24th and 28th weeks of gestation. Women with abnormal glucose levels ≥130 mg/dL (7.2 mmol/L) after 1 hour GCT underwent a standard 100 g 3 hour oral glucose tolerance test (OGTT) performed in the morning after eight hours overnight fasting. The diagnosis of GDM was confirmed if at least 2 of 4 glucose levels exceed Carpenter-Coustan criteria: fasting ≥ 95 mg/dL (5.3 mmol/L), 1 hour ≥ 180 mg/dL (10.0 mmol/L), 2 hours ≥ 155 mg/dL (8.6 mmol/L), and 3 hours ≥ 140 mg/dL (7.8 mmol/L).

Demographic and individual information such as maternal age, gestational week, parity were recorded. Weight and height of women with light clothes and without shoes were measured via a digital Seca Scale. BMI (Body Mass Index) was calculated by using the following formula: BMI=Weight (kg)/[Height (m) × Height (m)] and evaluated based on classification of (World Health Organisation) WHO as follows: >18.5 kg/m2 defined as underweight, 18.5-24.9 kg/m2 defined as normal weight range, 25.0-29.9 kg/m2 defined as overweight and ≥30.0 kg/m2 defined as obese. Investigators collected blood samples from each women between 24th and 28th weeks of pregnancy during their scheduled antenatal visit to determine the serum 25-hydroxyvitamin D [(25OHD)] concentration.

Levels of 25(OH)D on serum was measured by high performance liquid chromatography (HPLC) in biochemistry laboratory at Gulhane Education and Research Hospital. Investigators used clinical cutoffs based Institute of Medicine (IOM) criteria to categorize 25(OH)D levels: severe deficiency (<10 ng/mL), deficiency (10-20 ng/mL) and insufficiency (20-30 ng/mL).

Firstly, the variables were tested using Kolmogorov-Smirnov test to determine whether they are normally distributed. Descriptive analyses were presented as mean±standard deviation (SD) for normally distributed variables. Since the maternal age, serum 25(OH)D, log-transformed 50 g 1 hour GCT and log-transformed fasting blood glucose values were normally distributed; the Student's t-test was used to compare these parameters between women with and without GDM. Descriptive analyses were presented as median(min-max) for the non-normally distributed. Since the gestational age, gravity, and parity were not normally distributed; Mann-Whitney U test was used to compare these parameters between groups. Chi square test was used for categorical variable to compare the proportions in different groups. As both parameters were normally distributed, the correlation coefficients and their significance were calculated using the Pearson test. For the multivariate analysis, the possible factors identified with univariate analyses were further entered into the logistic regression analysis to determine independent predictors of women outcome. Hosmer-Lemeshow goodness of fit statistics were used to assess model fit. A 5% type-I error level was used to infer statistical significance. Receiver operating characteristics (ROC) analysis was done to identify the optimal cutoff point values of maternal serum 25OHD levels. All the data collected from the participants were analyzed using Statistical Package for the Social Sciences (SPSS) version 22.0 (SPSS Inc., Chicago, Illinois, USA) and p<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy,
* Aged in 20-40 years,
* Gestational age 24-28 weeks,
* Non-history of acute or chronic diseases.

Exclusion Criteria:

* History of GDM,
* Type 1 and 2 diabetes mellitus,
* Preeclampsia,
* Polycystic ovary syndrome,
* Thyroid disease
* Parathyroid disease,
* Metabolic bone disease,
* Kidney disease,
* Abnormal liver function,
* Multiple pregnancy, or
* Women receiving drugs related to calcium and vitamin D metabolism (with the exception of routine vitamin supplements prescribed during pregnancy)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In this observational cross-sectional study, 40 women with GDM and 40 healthy pregnant between 20-40 years in age, in their 24-28th gestational week applied to Gulhane Education and Research Hospital were recruited. This study must recruit 40 women for each group to have 80% study power with 5% type I error level to detect a clinically significant difference.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-01-05 (Actual); Primary Completion 2013-08-05 (Actual); Study Completion 2013-08-05 (Actual)

PRIMARY OUTCOMES:
Serum 25(OH)D levels | 24-28. weeks of pregnancy
  Levels of 25(OH)D on serum was measured by high performance liquid chromatography (HPLC) in biochemistry laboratory at Gulhane Education and Research Hospital.
Pre-pregnancy BMI | 24-28. weeks of pregnancy
  BMI (Body Mass Index) was calculated by using the following formula:
  BMI=Weight (kg)/[Height (m) × Height (m)].

CONTACTS AND LOCATIONS:
Overall Officials: Gülhan SAMUR, Professor, Principal Investigator — Hacettepe University; Gözde EDE, MSci, Study Chair — Hacettepe University; Müfit YENEN, Professor, Study Chair — Saglik Bilimleri Universitesi; Uğur KESKİN, Assoc. Prof., Study Chair — Gulhane Education and Research Hospital

REFERENCES:
- [Background] Kennelly MA, McAuliffe FM. Prediction and prevention of Gestational Diabetes: an update of recent literature. Eur J Obstet Gynecol Reprod Biol. 2016 Jul;202:92-8. doi: 10.1016/j.ejogrb.2016.03.032. Epub 2016 Apr 4. PMID 27235645
- [Background] Damm P, Houshmand-Oeregaard A, Kelstrup L, Lauenborg J, Mathiesen ER, Clausen TD. Gestational diabetes mellitus and long-term consequences for mother and offspring: a view from Denmark. Diabetologia. 2016 Jul;59(7):1396-1399. doi: 10.1007/s00125-016-3985-5. Epub 2016 May 12. PMID 27174368
- [Background] Zhang MX, Pan GT, Guo JF, Li BY, Qin LQ, Zhang ZL. Vitamin D Deficiency Increases the Risk of Gestational Diabetes Mellitus: A Meta-Analysis of Observational Studies. Nutrients. 2015 Oct 1;7(10):8366-75. doi: 10.3390/nu7105398. PMID 26437429
- [Background] Poel YH, Hummel P, Lips P, Stam F, van der Ploeg T, Simsek S. Vitamin D and gestational diabetes: a systematic review and meta-analysis. Eur J Intern Med. 2012 Jul;23(5):465-9. doi: 10.1016/j.ejim.2012.01.007. Epub 2012 Feb 21. PMID 22726378
- [Background] Burris HH, Rifas-Shiman SL, Kleinman K, Litonjua AA, Huh SY, Rich-Edwards JW, Camargo CA Jr, Gillman MW. Vitamin D deficiency in pregnancy and gestational diabetes mellitus. Am J Obstet Gynecol. 2012 Sep;207(3):182.e1-8. doi: 10.1016/j.ajog.2012.05.022. Epub 2012 Jun 1. PMID 22717271
- [Background] Mutlu N, Esra H, Begum A, Fatma D, Arzu Y, Yalcin H, Fatih K, Selahattin K. Relation of maternal vitamin D status with gestational diabetes mellitus and perinatal outcome. Afr Health Sci. 2015 Jun;15(2):523-31. doi: 10.4314/ahs.v15i2.27. PMID 26124799
- [Result] American Diabetes Association. Gestational diabetes mellitus. Diabetes Care. 2004 Jan;27 Suppl 1:S88-90. doi: 10.2337/diacare.27.2007.s88. No abstract available. PMID 14693936
- [Result] Wei SQ. Vitamin D and pregnancy outcomes. Curr Opin Obstet Gynecol. 2014 Dec;26(6):438-47. doi: 10.1097/GCO.0000000000000117. PMID 25310531
- [Result] Durnwald C. Gestational diabetes: Linking epidemiology, excessive gestational weight gain, adverse pregnancy outcomes, and future metabolic syndrome. Semin Perinatol. 2015 Jun;39(4):254-8. doi: 10.1053/j.semperi.2015.05.002. Epub 2015 Jun 17. PMID 26093518
- [Result] Sreelakshmi PR, Nair S, Soman B, Alex R, Vijayakumar K, Kutty VR. Maternal and neonatal outcomes of gestational diabetes: A retrospective cohort study from Southern India. J Family Med Prim Care. 2015 Jul-Sep;4(3):395-8. doi: 10.4103/2249-4863.161331. PMID 26288780
- [Result] Domaracki P, Sadlecki P, Odrowaz-Sypniewska G, Dzikowska E, Walentowicz P, Siodmiak J, Grabiec M, Walentowicz-Sadlecka M. Serum 25(OH) Vitamin D Levels in Polish Women during Pregnancies Complicated by Hypertensive Disorders and Gestational Diabetes. Int J Mol Sci. 2016 Sep 27;17(10):1574. doi: 10.3390/ijms17101574. PMID 27690002
- [Result] Lu M, Xu Y, Lv L, Zhang M. Association between vitamin D status and the risk of gestational diabetes mellitus: a meta-analysis. Arch Gynecol Obstet. 2016 May;293(5):959-66. doi: 10.1007/s00404-016-4010-4. Epub 2016 Jan 29. PMID 26825733
- [Result] Pirjani R, Shirzad N, Qorbani M, Phelpheli M, Nasli-Esfahani E, Bandarian F, Hemmatabadi M. Gestational diabetes mellitus its association with obesity: a prospective cohort study. Eat Weight Disord. 2017 Sep;22(3):445-450. doi: 10.1007/s40519-016-0332-2. Epub 2016 Oct 17. PMID 27747467
- [Result] Jelsma JG, van Poppel MN, Galjaard S, Desoye G, Corcoy R, Devlieger R, van Assche A, Timmerman D, Jans G, Harreiter J, Kautzky-Willer A, Damm P, Mathiesen ER, Jensen DM, Andersen L, Dunne F, Lapolla A, Di Cianni G, Bertolotto A, Wender-Oegowska E, Zawiejska A, Blumska K, Hill D, Rebollo P, Snoek FJ, Simmons D. DALI: Vitamin D and lifestyle intervention for gestational diabetes mellitus (GDM) prevention: an European multicentre, randomised trial - study protocol. BMC Pregnancy Childbirth. 2013 Jul 5;13:142. doi: 10.1186/1471-2393-13-142. PMID 23829946